CLINICAL TRIAL: NCT03564327
Title: Clinical Prognosis of Patients With Atrial Fibrillation During Radiofrequency Ablation and Interest of the Isochron Map
Brief Title: Clinical Prognosis of Patients With Atrial Fibrillation During Radiofrequency Ablation
Acronym: Isochrone-AFAn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-03/MG-02
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with atrial fibrillation (Experimental)
  Interventions: Procedure: External electric cardioversion

INTERVENTIONS:
Procedure: External electric cardioversion — Three attempts (200-250 joules)

SUMMARY:
Identify the parameters of the predictive isochronous map for the clinical outcome of radiofrequency ablation in terms of absence of documented atrial fibrillation recurrence at 18 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient is available for 18 month follow-up
* The patient has paroxysmal or persistent atrial fibrillation

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding Early Study Exit Criteria: Patient does not have paroxysmal or persistent AF at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation relapse in non-reducible or non-inducible patients | Month 18
  Atrial fibrillation detected by routine or event-associated Holter examination

SECONDARY OUTCOMES:
Atrial fibrillation relapse in non-reducible or non-inducible patients | Month 12
  Atrial fibrillation detected by routine or event-associated Holter examination
Arrhythmia occurrence in non-reducible or non-inducible patients | Month 12
  Arrhythmia, including atrial tachycardia detected by routine or event-associated Holter examination
Arrhythmia occurrence in non-reducible or non-inducible patients | Month 18
  Arrhythmia, including atrial tachycardia detected by routine or event-associated Holter examination
Identification of zones of low voltage on voltage maps in non-inducible patients | Day 0
  Yes/No
Identification of zones of anisochronic zones on voltage maps in non-inducible patients | Day 0
  Yes/No
Maximum variation of conduction speed in the same anatomic region in non-inducible patients | Day 0
  %
Decreasing velocities in the same anatomic region in non-inducible patients | Day 0
  %
Wave front rotation in the same anatomic region in non-inducible patients | Day 0
  degrees
Total time of radiofrequency in non-inducible patients | Day 0
  Minutes
Total procedure time in non-inducible patients | Day 0
  Minutes
Comparison of lesion volume in non-inducible patients | Day 0
  Force-time integral, lesion size index or stroke volume index
Number and size of treated zones by guided versus conventional ablation in non-inducible patients | Day 0
  cm2
List locations most frequently treated | Day 0
  Number of each
Survival without relapse of patients treated using the Carto- vs Rhythmia-guided ablation approaches in non-reducible or non-inducible patients | Month 18
  Atrial fibrillation detected by routine or event-associated Holter examination
Arrhythmia occurrence in non-reducible or non-inducible patients | Month 18
  Atrial fibrillation detected by routine or event-associated Holter examination

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Granier, MD, Principal Investigator — CHU de Montpellier
Locations (2):
- France (2):
  - CHU Montpellier, Montpellier
  - CHU Nimes, Nîmes